CLINICAL TRIAL: NCT07174362
Title: QUAD-HF Registry - A Prospective Registry of Patients With Incident Heart Failure and Left Ventricular Ejection Fraction of <50%
Brief Title: QUAD-HF - Prospective Registry of Patients With Incident Heart Failure and Left Ventricular Ejection Fraction <50%
Acronym: QUAD-HF
Status: Recruiting | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other); British Society for Heart Failure (Unknown)
Responsible Party: Sponsor
Other Study IDs: 354730
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Observational Cohort; Heart Failure; Longitudinal
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The QUAD-HF registry is an observational study that would enroll patients in the United Kingdom, who have been newly diagnosed with heart failure and a left ventricular ejection fraction <50%. We plan to assess clinical outcomes in these patients, such as hospitalization and death, in relation to their diagnosis, implementation of guidelines and type of treatments these patients have received.

DETAILED DESCRIPTION:
Heart failure (HF) is a widespread global health challenge, affecting approximately 1 million individuals in the United Kingdom and the prevalence is predicted to almost double in the next decades due to the ageing population. In the United Kingdom, hospitalizations for HF account for 5% of emergency medical admissions with a substantial economic burden.

The management of heart failure however is a true success story of modern medicine. Four decades of randomised clinical trials, provide the evidence base for an extensive catalogue of disease-modifying pharmacological and device treatments that have improved prognosis, particularly in patients with HF and a reduced LVEF <50%.

However, controlled studies tend to evaluate treatments in selected patient cohorts defined by strict trial inclusion criteria and often exclude older patients, include less women and patient background is often non-diverse. Furthermore, while within clinical trials these treatments are readily available and delivered to patients in meticulous and tightly controlled settings, this does not usually reflect real-world clinical environments, where there may be resource deficiencies. Indeed, a recent cross-sectional survey of hospital-based HF services in the UK, demonstrates wide variation in access to treatment and services. It is therefore important to evaluate the utilization of these treatments and adherence to practice guidelines in a real-world setting.

In England & Wales, a National Heart Failure Audit collects data in patients with HF who have unplanned hospitalisations for worsening symptoms. This does not extend outside of hospital settings, where the majority of patients time is spent managing their condition. The UK HFpEF study is an ongoing study which caters for patients who have heart failure with a preserved left ventricular ejection fraction (>50%).

There is however no readily available database or registry outside of hospital, that provides contemporaneous information about the care, changes in management or long-term outcomes for patients with HF and a left ventricular ejection fraction of <50%, as exists in other healthcare systems.

The QUAD-HF registry is designed as a UK multi-centre, prospective longitudinal registry and would enrol adult patients (>18 years) who present with incident heart failure and a left ventricular ejection fraction <50%. NHS secondary or primary care centres in the United Kingdom would be invited to enroll patients into the registry if they have an established HF clinic that routinely documents patient characteristics and pharmacological therapy at each visit. Site selection would be by the steering committee.

Consecutive ambulatory patients attending these clinics, would be approached by managing clinicians; usually specialist HF nurses or cardiologists; to participate. For those hospitalized at the time of their new diagnosis, this approach would be by treating clinician when they are clinically stable. All patients would be treated according to contemporary guidelines.

In the initial phase of the study (1st 12 months), investigators aim to recruit 10 sites, with each site expected to enroll 100 patients into the study over 18 months. Additional sites will be invited as the registry develops. Selection of sites will be determined by the Steering Committee. At that recruitment rate and with additional sites added, investigators expect to onboard approximately 4000 participants into the registry by month 60.

Participants will provide oral and written informed consent to enable future data linkage of data relevant to their past and future health from medical, health, social care and other health-related records, which are collected or held in local, regional and national systems. The study has received ethical approval from the Cambridgeshire South Research Ethics Committee (25/EE/0088) and local research and development departments of participating hospitals.

Broadly, the registry will evaluate the implementation of current HF guidelines and assess the quality of care in daily clinical practice in these patients. The primary clinical endpoint is a composite of cardiovascular mortality and hospitalization for heart failure, 1 year after diagnosis. Secondary endpoints include components of the primary endpoint, all-cause mortality, QUAD score at final therapy titration, days alive out of hospital, time to first HF-related hospitalization and patient-reported outcome measures.

The QUAD-HF registry would provide longitudinal analysis of profiles, management and outcomes for patients with incident HF and a left ventricular ejection fraction of <50% and provide a platform to support improved knowledge, the development of personalized care and support future research for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Newly diagnosed Heart Failure with a Left Ventricular Ejection Fraction <50% (≤12 Weeks prior to enrolment).
3. Able and willing to consent.

Exclusion Criteria:

1. LVEF 50% or more at time of diagnosis
2. Palliative care
3. Unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants would include adult patients (>18 years) attending HF clinics in hospital or community settings or those hospitalized for the management of Acute Decompensated Heart failure (ADHF), who have been newly diagnosed HF with a left ventricular ejection fraction of <50%, no more than 12 weeks prior. Patients would be excluded if they have had a previous diagnosis of heart failure, are on a palliative care pathway or are unable or unwilling to consent.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Mortality or Hospitalization for Heart Failure | From enrolment to 12 months after diagnosis
  Death due to cardiac causes or hospitalization due to worsening heart failure symptoms

SECONDARY OUTCOMES:
All-cause mortality | From enrolment to 12 months after diagnosis
  Death due to any cause
Cardiovascular Mortality | From enrolment to 12 months after diagnosis
  Death due to cardiac causes
Hospitalization for Heart Failure | From enrolment to 12 months after diagnosis
  Hospitalization due to worsening heart failure symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Henry Oluwasefunmi Savage, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Mid and South Essex NHS Foundation Trust, Basildon, Essex
  - British Heart Foundation Glasgow Cardiovascular Research Centre, Glasgow, Glasgow

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data from this study cannot be shared publicly, or outside the United Kingdom, due to the restrictions of ethical approval obtained, internal regulations, patient consent, and data regulations. Researchers from within the United Kingdom will require approval from the executive steering committee of the registry, for IPD to be made available. Researchers from outside the United Kingdom interested in collaboration are invited to contact the principal investigator to discuss.

REFERENCES:
- [Background] UK HFpEF Collaborative Group. Rationale and design of the United Kingdom Heart Failure with Preserved Ejection Fraction Registry. Heart. 2024 Feb 12;110(5):359-365. doi: 10.1136/heartjnl-2023-323049. PMID 37827557
- [Background] National Institute for Cardiovascular Outcomes Research (NICOR). https://www.nicor.org.uk/~documents/route%3A/download/2765. 2024 [cited 2025 Jan 30]. National Heart failure Audit (NHFA) 2024 Summary Report.
- [Background] Nallamothu BK, Hayward RA, Bates ER. Beyond the randomized clinical trial: the role of effectiveness studies in evaluating cardiovascular therapies. Circulation. 2008 Sep 16;118(12):1294-303. doi: 10.1161/CIRCULATIONAHA.107.703579. No abstract available. PMID 18794402
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- See also: Health Research Authority, Research Summary Page — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/quad-hf-registry/